CLINICAL TRIAL: NCT04312802
Title: Measurement of Cardiopulmonary Exercise Capacity in Patients with Type 1 Diabetes Mellitus Approaching Simultaneous Kidney Pancreas Transplantation
Brief Title: Cardiopulmonary Testing for Potential Pancreas Transplant Candidates
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Edward Sharples, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 251119v1.1
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Risk Factor; Diabetes Mellitus, Type 1; Pancreas Transplant; Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Single arm observational study
  Interventions: Diagnostic Test: Cardiopulmonary exercise test (CPET)

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test (CPET) — The participant will undergo a cardio-pulmonary exercise test (CPET) on a cycle ergometer (Ergoline) connected to a 12-lead electrocardiogram, oxygen saturation monitor and continuous non-invasive blood pressure cuff. Respiratory gas exchanged will be measured from a tight fitting facemask. An initial 2-min period of baseline data will be collected at rest before a 180-s period of unloaded cycling. A ramp protocol will then be applied and the participant will be instructed to continue cycling at a constant cadence of 60 rpm as long as they can. The test will be terminated if the participant indicates that:
  * they cannot continue
  * cadence falls to <55 rpm due to fatigue or dyspnoea
  * they develop abnormal cardiac signs or symptoms, such as ischaemia and arrhythmia.

SUMMARY:
Patients being assessed for Kidney Pancreas transplantation often have pre-existing co-morbid disease that contributes to structural cardiac and vascular disease. There is no consensus on optimal pre-listing cardiac assessment to reliably minimize risk of peri-operative cardiac events. Functional status using the cardio-pulmonary exercise test (CPET) has been used in cardiac and abdominal surgery, including abdominal aortic aneurysm (AAA) repair and kidney transplantation, but high risk patients with diabetes are often lacking from these studies. This study will investigate the correlation between function, measures using CPET and standard cardiac assessment, and determine the variation in usual measures of anaerobic threshold and VO2 max in this population.

DETAILED DESCRIPTION:
20 participants will be recruited to a blinded observational study. Patients referred for pancreas kidney transplantation assessment will be provided information about the study. They will subsequently be approached at their initial assessment visit and informed consent will be taken.

Participants will have standard clinical assessment which includes:

1. Clinical history and examination
2. 12 lead electrocardiogram (ECG)
3. Chest X-ray (CXR)
4. Myocardial perfusion imaging (MPS)
5. If MPS imaging is suggestive of stress induced ischaemia, or severe left ventricular (LV) dysfunction, the participant will undergo coronary angiography as part of standard assessment protocol.

In addition, study participants will undergo CPET testing. This will take place within 1 week of the standard peri-operative cardiac assessment. The results of this investigation will be recorded against a unique identifier on a secure Oxford University Hospital computer. Information about the study or participants' individual results will not normally be disclosed to the participant or clinical team, and so will not influence clinical management. However if, when the results are analysed, the research team note a CPET result that suggests a clear and significant impairment of functional reserve such that the participant should not be listed, this result will be disclosed to the individual and their medical team so that the information can be used in order to make the safest decision about transplant listing. There will be no further clinical visits but participants will consent to collection of their clinical data until 3 months post-transplant, or until they are removed from the waiting list.

At the end of the study, the results of CPET testing will be correlated to measures from standard cardiac investigations and to peri-operative cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent
* Diagnosed with type 1 diabetes mellitus with estimated glomerular filtration rate (eGFR)<20ml/min or on renal replacement therapy referred for simultaneous pancreas-kidney (SPK) transplant

Exclusion Criteria:

* Participant unable to undergo CPET testing due to limitation on mobility or limb movement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with type 1 diabetes mellitus and impaired kidney function being assessed for simultaneous kidney pancreas transplantation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Anaerobic threshold (AT) measurement correlation with cardiac perfusion | Single 1 day test
  Comparison of AT measurement and MPS imaging result

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sharples, MBBS PhD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No